CLINICAL TRIAL: NCT06919185
Title: Short- and Long-term Effects of Robot-assisted Plication in Diaphragmatic Paralysis - the Prospective RAPIDLY-study
Brief Title: Short- and Long-term Effects of Robot-assisted Plication in Diaphragmatic Paralysis
Acronym: RAPIDLY
Status: Not yet recruiting | Type: Observational
Sponsor: Uppsala County Council, Sweden (Other Government)
Collaborators: Uppsala University (Other)
Responsible Party: Principal Investigator, Andreas Palm, Associate Professor, Uppsala County Council, Sweden
Other Study IDs: 2025-01028-01
Record Dates: First submitted 2025-03-26; First posted 2025-04-09 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Diaphragmatic Plication; Diaphragmatic Paralysis; Diaphragmatic Eventration
Keywords: RATS; robot-assisted thoracic surgery; plication; dyspnea; thoracotomy
MeSH Terms: conditions — Respiratory Paralysis; Diaphragmatic Eventration; Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients accepted for Robot-assisted diaphragmatic plication: Patients with symptomatic unilateral diaphragmatic paralysis persisting for ≥1 year accepted for Robot-assisted diaphragmatic plication at 5 Swedish University Hospitals, Gothenburg, Linköping, Lund, Umeå, and Uppsala

SUMMARY:
Diaphragmatic paralysis may lead to severe symptoms such as breathlessness and reduced physical capacity.

Diaphragmatic plication using Robotic-Assisted Thoracic Surgery (RATS) is a minimally invasive surgical technique developed to improve lung function by correcting diaphragmatic elevation.

While its benefits have been reported in retrospective reports, prospective studies are lacking.

This prospective observational cohort study aimsto evaluate the short- and long-term effects of robot-assisted diaphragmatic plication on subjective breathlessness, physical performance, lung function, blood gases, and imaging findings at five Swedish university hospitals: Gothenburg, Linköping, Lund, Umeå, and Uppsala.

Patients will be assessed preoperatively and postoperatively after one to three months and after one and three years.

DETAILED DESCRIPTION:
Assessments

Patient characteristics:

Age, sex, height, and weight will be recorded. Body mass index (BMI) is calculated by dividing a person's weight by their height in meters squared.

Aetiology of diaphragmatic paralysis, relevant co-morbidities and use of long-term oxygen therapy and/or mechanical ventilation will be recorded.

The date for symptom debut, if known, is recorded. Smoking history is defined as current smoker, ex-smoker (smoking history of ≥100 cigarettes and having quit smoking ≥6 months ago), and never smoker (smoking history of <100 cigarettes). Smoking is quantified by pack-years (the number of packs of cigarettes a person has smoked daily, multiplied by the number of years they have smoked).

Primary outcome:

The patients' exercise capacity will be evaluated using the 6-minute walking distance (6MWD). The patients are asked to walk as far as possible on a flat, straight surface for six minutes, and the total distance walked is measured.

Secondary outcomes:

Questionnaires:

The modified Borg Scale is a tool with a range from 0 to 10 used to measure an individual's perceived level of breathlessness or muscle fatigue during physical activity, where 0 represents no breathlessness, and 10 represents maximal breathlessness.

The modified Medical Research Council (mMRC) dyspnea scale is used to assess the severity of breathlessness. The scale ranges from 0 to 4, with higher scores indicating more significant breathlessness.

The Dyspnea-12 is a questionnaire used to measure the severity and quality of breathlessness in individuals with respiratory or cardiovascular conditions. It assesses dyspnea's physical and emotional aspects, providing a comprehensive picture of how breathlessness affects a person's life. It consists of 12 items, each with a scale range between 0 (no dyspnea) and 3 (severe dyspnea).

The EuroQol-5-dimension (EQ-5D) questionnaire is one of the most widely used tools for assessing health-related quality of life. It includes five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. These dimensions create a descriptive profile that can be converted into a single summary index, where a score of 1.0 indicates perfect health. Additionally, the tool includes a Visual Analog Scale (VAS), ranging from 0 (worst imaginable health) to 100 (best imaginable health), for self-assessment of overall health status.

Spirometry Spirometry will be conducted 15 minutes after bronchodilation (inhalation of 200 µg salbutamol) in both supine and upright positions. Body plethysmography and single-breath Diffusing Capacity in the Lungs for Carbon Monoxide (DLCO) measurement will be performed. Predicted values will be determined using reference equations from the Global Lung Function Initiative (GLI).

One-minute sit-to-stand test (1-MSTST) This test assesses a person's functional exercise capacity by recording the number of full sit-to-stand repetitions completed in 60 seconds.

The Maximal Inspiratory Pressure (MIP) test is a respiratory test that measures the strength of the inspiratory muscles, particularly the diaphragm. By inhaling as forcefully as possible in a handheld device, the maximum negative pressure generated is recorded.

Blood gas analysis A capillary or arterial blood gas analysis obtains the partial pressure of oxýgen and carbon dioxide (PaCO2) in kilo Pascal (kPa) and Base Excess (BE) in mmol/l. Pulse oximetry obtains oxygen saturation.

Chest X-ray Chest X-rays are acquired in full inspiration and expiration in frontal and lateral views. The distance from the most cranial part of the lung to the highest part of the diaphragm in both frontal and side views are measured separately.

Computerised tomography (CT) of Thorax A CT with a standard protocol to identify and quantify lower lobe atelectasis.

Adverse events Operating time, chest-drain duration, length of hospitalisation, per- and postoperative complications such as pain, bleeding and infections, 30-day readmission and 30-days mortality are recorded.

Statistics Descriptive statistics summarise the data, and inferential statistics compare group differences.

Associations with the outcomes will be analysed using multivariable regression models, including linear regression (for continuous outcome variables) and logistic regression (for categorical outcomes). Repeated measurements within individuals will be managed through multilevel, random-effects models.

Power calculation: Based on a standard deviation of 90 meters in the 6-minute walk test (6MWT) among the general population, and considering that the minimal clinically important difference (MCID) is 53 meters, a total of 45 patients is required.

Assessments pre-operatively Demographics Anthropometrics Co-morbidities Questionnaires Physical capacity tests Spirometry MIP Blood gas analysis Chest X-ray CT scan

Assessments 1-3 months post-operatively Anthropometrics Questionnaires Physical capacity tests Spirometry MIP Blood gas analysis Chest X-ray CT scan

Assessments after 1 and 3 years post-operatively Anthropometrics Questionnaires Physical capacity tests Spirometry MIP Blood gas analysis Chest X-ray

Ethical considerations:

Robot-assisted diaphragm plication is performed at several university hospitals in Sweden and abroad. The patients in this study have been clinically approved for this surgery. They are not exposed to any additional risks in this study beyond being examined more thoroughly with surveys and questionnaires, lung function and performance tests, and chest X-rays before and after the surgical procedure. The study is approved by the Swedish Ethical Review Authority, Dnr 2025-01028-01.

Relevance of research:

Robot-assisted plication in diaphragmatic paralysis is a new operative method performed at many thoracic centres worldwide without being scientifically evaluated in prospective studies. This national multicenter study, with a large cohort by international standards and with validated, highly relevant outcome variables, is expected to gain significant attention among thoracic surgeons and pulmonary physicians worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic unilateral diaphragmatic paralysis persisting for ≥1 year
* Patients are scheduled for RATS at thoracic surgery clinics in five Swedish university hospitals (Gothenburg, Linköping, Lund, Umeå, and Uppsala).

Exclusion Criteria:

* Inability to complete forms in Swedish
* Neuromuscular disease as the cause of diaphragmatic paralysis
* Other significant causes of dyspnea
* Impaired physical capacity from other causes than diaphragmatic paralysis.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unilateral diaphragmatic paralysis
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2031-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
6-minute walking distance (6MWD). | From enrollment to end of observation att 3 years.
  The patients are asked to walk as far as possible on a flat, straight surface for six minutes, and the total distance walked is measured.

SECONDARY OUTCOMES:
The modified Borg Scale | From enrollment to end of observation att 3 years.
  A tool with a range from 0 to 10 used to measure an individual's perceived level of breathlessness or muscle fatigue during physical activity, where 0 represents no breathlessness, and 10 represents maximal breathlessness
The modified Medical Research Council (mMRC) dyspnea scale | From enrollment to end of observation att 3 years.
  The mMRC is used to assess the severity of breathlessness. The scale ranges from 0 to 4, with higher scores indicating more significant breathlessness
The Dyspnea-12 questionnaire | From enrollment to end of observation att 3 years.
  The Dyspnea-12questionnaire is used to measure the severity and quality of breathlessness in individuals with respiratory or cardiovascular conditions. It assesses dyspnea's physical and emotional aspects, providing a comprehensive picture of how breathlessness affects a person's life. It consists of 12 items, each with a scale range between 0 (no dyspnea) and 3 (severe dyspnea)
The EQ-5D questionnaire | From enrollment to end of observation att 3 years.
  The EQ-5D is one of the most widely used tools for assessing health-related quality of life. It includes five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. These dimensions create a descriptive profile that can be converted into a single summary index, where a score of 1.0 indicates perfect health. Additionally, the tool includes a Visual Analog Scale (VAS), ranging from 0 (worst imaginable health) to 100 (best imaginable health), for self-assessment of overall health status
Spirometry | From enrollment to end of observation att 3 years.
  Spirometry will be conducted 15 minutes after bronchodilation (inhalation of 200 µg salbutamol) in both supine and upright positions. Body plethysmography and single-breath DLCO measurement will be performed. Predicted values will be determined using reference equations from the Global Lung Function Initiative
One-minute sit-to-stand test (1-MSTST) | From enrollment to end of observation att 3 years.
  This test assesses a person's functional exercise capacity by recording the number of full sit-to-stand repetitions completed in 60 seconds
The Maximal Inspiratory Pressure (MIP) test | From enrollment to end of observation att 3 years.
  MIP is a respiratory test that measures the strength of the inspiratory muscles, particularly the diaphragm. By inhaling as forcefully as possible in a handheld device, the maximum negative pressure generated is recorded
Blood gas analysis | From enrollment to end of observation att 3 years.
  A capillary or arterial blood gas analysis obtains the partial pressure of oxýgen (O2).
Blood gas analysis | From enrollment to end of observation att 3 years.
  A capillary or arterial blood gas analysis obtains the partial pressure of carbon dioxide (CO2)
Blood gas analysis | From enrollment to end of observation att 3 years.
  A capillary or arterial blood gas analysis obtains the levels of base excess (BE)
Pulse oximetry | From enrollment to end of observation att 3 years.
  Obtains oxygen saturation.
Chest X-ray | From enrollment to end of observation att 3 years.
  Chest X-rays are acquired in full inspiration and expiration in frontal and lateral views. The distance from the most cranial part of the lung to the highest part of the diaphragm in both frontal and side views are measured separately.
Computerised tomography (CT) of Thorax | From enrollment to end of observation att 3 years.
  A CT with a standard protocol to identify and quantify lower lobe atelectasis.
Adverse events | 30 days post-operatively
  Operating time, chest-drain duration, length of hospitalisation, per- and postoperative complications such as pain, bleeding and infections, 30-day readmission and 30-days mortality are recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Palm, Md, PhD, Principal Investigator — Uppsala University Hospital
Locations (1):
- Department of Medical Sciences, Lung-, Allergy-, and Sleep Research, Uppsala University/Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No
Individual Partisipant Data (IPD) can be shared after an application to the Swedish Ethics Review Authority has been accepted.

REFERENCES:
- [Background] Marmor HN, Xiao D, Godfrey CM, Nesbitt JC, Gillaspie EA, Lambright ES, Bacchetta M, Moe DM, Deppen SA, Grogan EL. Short-term outcomes of robotic-assisted transthoracic diaphragmatic plication. J Thorac Dis. 2023 Apr 28;15(4):1605-1613. doi: 10.21037/jtd-22-442. Epub 2023 Mar 28. PMID 37197490
- [Background] Crook S, Busching G, Schultz K, Lehbert N, Jelusic D, Keusch S, Wittmann M, Schuler M, Radtke T, Frey M, Turk A, Puhan MA, Frei A. A multicentre validation of the 1-min sit-to-stand test in patients with COPD. Eur Respir J. 2017 Mar 2;49(3):1601871. doi: 10.1183/13993003.01871-2016. Print 2017 Mar. PMID 28254766
- [Background] Quanjer PH, Stanojevic S, Cole TJ, Baur X, Hall GL, Culver BH, Enright PL, Hankinson JL, Ip MS, Zheng J, Stocks J; ERS Global Lung Function Initiative. Multi-ethnic reference values for spirometry for the 3-95-yr age range: the global lung function 2012 equations. Eur Respir J. 2012 Dec;40(6):1324-43. doi: 10.1183/09031936.00080312. Epub 2012 Jun 27. PMID 22743675
- [Background] Dolan P. Modeling valuations for EuroQol health states. Med Care. 1997 Nov;35(11):1095-108. doi: 10.1097/00005650-199711000-00002. PMID 9366889
- [Background] Yorke J, Moosavi SH, Shuldham C, Jones PW. Quantification of dyspnoea using descriptors: development and initial testing of the Dyspnoea-12. Thorax. 2010 Jan;65(1):21-6. doi: 10.1136/thx.2009.118521. Epub 2009 Dec 8. PMID 19996336
- [Background] Olsson M, Ekstrom M. Validation of the Dyspnoea-12 and Multidimensional Dyspnea profile among older Swedish men in the population. BMC Geriatr. 2022 Jun 2;22(1):477. doi: 10.1186/s12877-022-03166-5. PMID 35655151
- [Background] Munari AB, Gulart AA, Dos Santos K, Venancio RS, Karloh M, Mayer AF. Modified Medical Research Council Dyspnea Scale in GOLD Classification Better Reflects Physical Activities of Daily Living. Respir Care. 2018 Jan;63(1):77-85. doi: 10.4187/respcare.05636. Epub 2017 Sep 5. PMID 28874609
- [Background] Holland AE, Spruit MA, Troosters T, Puhan MA, Pepin V, Saey D, McCormack MC, Carlin BW, Sciurba FC, Pitta F, Wanger J, MacIntyre N, Kaminsky DA, Culver BH, Revill SM, Hernandes NA, Andrianopoulos V, Camillo CA, Mitchell KE, Lee AL, Hill CJ, Singh SJ. An official European Respiratory Society/American Thoracic Society technical standard: field walking tests in chronic respiratory disease. Eur Respir J. 2014 Dec;44(6):1428-46. doi: 10.1183/09031936.00150314. Epub 2014 Oct 30. PMID 25359355
- [Background] Casanova C, Celli BR, Barria P, Casas A, Cote C, de Torres JP, Jardim J, Lopez MV, Marin JM, Montes de Oca M, Pinto-Plata V, Aguirre-Jaime A; Six Minute Walk Distance Project (ALAT). The 6-min walk distance in healthy subjects: reference standards from seven countries. Eur Respir J. 2011 Jan;37(1):150-6. doi: 10.1183/09031936.00194909. Epub 2010 Jun 4. PMID 20525717
- [Background] Ekstrom M, Li PZ, Lewthwaite H, Bourbeau J, Tan WC, Jensen D. The modified Borg/6-min walk distance ratio: a method to assess exertional breathlessness and leg discomfort using the 6-min walk test. ERJ Open Res. 2023 Sep 25;9(5):00281-2023. doi: 10.1183/23120541.00281-2023. eCollection 2023 Sep. PMID 37753276
- [Background] Burns DM. Epidemiology of smoking-induced cardiovascular disease. Prog Cardiovasc Dis. 2003 Jul-Aug;46(1):11-29. doi: 10.1016/s0033-0620(03)00079-3. PMID 12920698
- [Background] Hunt AR, Stuart CM, Gergen AK, Bang TJ, Reihman AE, Helmkamp LJ, Lin Y, Mitchell JD, Meguid RA, Scott CD, Wojcik BM. Long-Term Patient-Reported Symptom Improvement and Quality of Life after Transthoracic Diaphragm Plication in Adults. J Am Coll Surg. 2023 Sep 1;237(3):533-544. doi: 10.1097/XCS.0000000000000762. Epub 2023 May 17. PMID 37194947
- [Background] Le UT, Titze L, Hundeshagen P, Passlick B, Schmid S. Robotic diaphragm plication: functional and surgical outcomes of a single-center experience. Surg Endosc. 2023 Jun;37(6):4795-4802. doi: 10.1007/s00464-023-09942-7. Epub 2023 Mar 13. PMID 36914782
- [Background] Lampridis S, Pradeep IHDS, Bille A. Robotic-assisted diaphragmatic plication: Improving safety and effectiveness in the treatment of diaphragmatic paralysis. Int J Med Robot. 2022 Jun;18(3):e2368. doi: 10.1002/rcs.2368. Epub 2022 Jan 24. PMID 35041770
- [Background] Valenti J, Tan K, Rubino K, Hanhan Z, Vega D, Kaufman M, Bauer T. Quality-of-life impact of diaphragm plication in patients with diaphragmatic paralysis: A retrospective study. Ann Thorac Med. 2024 Jan-Mar;19(1):105-111. doi: 10.4103/atm.atm_158_23. Epub 2024 Jan 25. PMID 38444988
- [Background] Zwischenberger BA, Kister N, Zwischenberger JB, Martin JT. Laparoscopic Robot-Assisted Diaphragm Plication. Ann Thorac Surg. 2016 Jan;101(1):369-71. doi: 10.1016/j.athoracsur.2015.05.118. PMID 26694286
- [Background] Kosse NJ, Galetin T, Schwarz SB, Mathes T, Koryllos A, Lopez-Pastorini A, Beckers F, Stoelben E. Results of the Diaphragmatic Plication Database: 10 Years' Experience. Thorac Cardiovasc Surg. 2023 Sep;71(6):483-489. doi: 10.1055/s-0041-1735496. Epub 2021 Oct 15. PMID 34655069
- [Background] Freeman RK, Van Woerkom J, Vyverberg A, Ascioti AJ. Long-term follow-up of the functional and physiologic results of diaphragm plication in adults with unilateral diaphragm paralysis. Ann Thorac Surg. 2009 Oct;88(4):1112-7. doi: 10.1016/j.athoracsur.2009.05.027. PMID 19766791
- [Background] Beshay M, Abdel Bary M, Kosek V, Vordemvenne T, Mertzlufft F, Schulte Am Esch J. Minimally-Invasive Diaphragmatic Plication in Patients with Unilateral Diaphragmatic Paralysis. J Clin Med. 2023 Aug 15;12(16):5301. doi: 10.3390/jcm12165301. PMID 37629343
- [Background] Gharagozloo F, McReynolds SD, Snyder L. Thoracoscopic plication of the diaphragm. Surg Endosc. 1995 Nov;9(11):1204-6. doi: 10.1007/BF00210929. PMID 8553235
- [Background] Freeman RK, Wozniak TC, Fitzgerald EB. Functional and physiologic results of video-assisted thoracoscopic diaphragm plication in adult patients with unilateral diaphragm paralysis. Ann Thorac Surg. 2006 May;81(5):1853-7; discussion 1857. doi: 10.1016/j.athoracsur.2005.11.068. PMID 16631685
- [Background] Gazala S, Hunt I, Bedard EL. Diaphragmatic plication offers functional improvement in dyspnoea and better pulmonary function with low morbidity. Interact Cardiovasc Thorac Surg. 2012 Sep;15(3):505-8. doi: 10.1093/icvts/ivs238. Epub 2012 Jun 12. PMID 22691375
- See also: Brief information about the study on Swedish Respiratory Society´s website — https://slmf.se/forskning/lungmedicinsk-forskning/sparc/
- Available data/document: Study Protocol: 2025-01028-01 — https://slmf.se/forskning/lungmedicinsk-forskning/sparc/

DOCUMENTS (1):
  • Study Protocol (2025-04-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT06919185/Prot_000.pdf